CLINICAL TRIAL: NCT01636037
Title: Augmentation of Antipsychotics With L-Dopa (Sinemet)
Brief Title: Antipsychotic Augmentation With L-Dopa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, George Foussias, Sub-Investigator, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156/2011
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; negative symptoms; deficit syndrome; SANS; Sinemet; L-dopa; levodopa; carbidopa; augmentation; antipsychotics
MeSH Terms: conditions — Schizophrenia | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-Dopa (Sinemet) (Experimental): Augmentation of current antipsychotic treatment with oral L-Dopa (levodopa/carbidopa) up to 900mg daily for 8 weeks
  Interventions: Drug: levodopa/carbidopa (generic version of Sinemet)

INTERVENTIONS:
Drug: levodopa/carbidopa (generic version of Sinemet) — Oral levodopa 900mg daily as tolerated.
  Other Names: Levodopa/carbidopa; Sinemet

SUMMARY:
Dopamine, a chemical in the brain, has been linked to schizophrenia for a number of years. More recently, there is evidence that certain areas affected in schizophrenia (e.g. motivation, cognition) may reflect too little dopamine, whereas symptoms like hallucinations and delusions have been linked to too much dopamine.

This study is designed to evaluate the safety, tolerability, and efficacy of giving L-dopa (Sinemet) to see if it will improve those symptoms related to too little dopamine. L-dopa has been approved for other medical conditions (e.g. Parkinson's disease) and works to increase levels of dopamine.

The investigators are linking this study with neuroimaging (fMRI) which will allows us to link any changes the investigators might find in clinical symptoms with changes in the brain. This information can prove useful in better understanding the mechanisms that account for these symptoms, as well as possible new treatments.

At present , treatments for these other symptoms that seem important in functional measures of outcome (i.e. deficit symptoms, including amotivation; cognitive symptoms) in schizophrenia have not proven particularly effective. It is hoped that L-dopa may provide a treatment that is more effective; going forward, this information would also be useful in drug development and future lines of investigation.

1. L-dopa will prove effective in improving deficit (also called 'primary negative' e.g. amotivation) and cognitive symptoms in schizophrenia.
2. It will be well tolerated and not increase risk of psychotic symptoms when administered in conjunction with their regular antipsychotic medications.

DETAILED DESCRIPTION:
Pharmacological (and non-pharmacological) strategies that may significantly improve the negative and cognitive symptoms of schizophrenia represent a critical unmet therapeutic need. There is wide acceptance of the notion that both negative and cognitive symptoms are best understood as features of hypo- rather than hyperdopaminergic activity. The primary negative and cognitive symptoms appear central to schizophrenia and predate the neurodevelopmental changes that subsequently give rise to the hyperdopaminergic state underlying positive symptoms. In using L-Dopa specifically, we avoid the abuse potential of agents such as the psychostimulants, or perturbations in pharmacological action as a function of dose, as observed with dopamine agonists. Further, more recent neuroimaging studies have provided in vivo evidence in keeping with the underlying rationale. First, imaging studies have demonstrated that L-dopa induces shifts in activity in both cortical and subcortical structures linked to reward, affect and cognition. Along similar lines, L-dopa-induced changes have been associated with improvement in motivation, cognitive tasks, and affect.

ELIGIBILITY:
Inclusion Criteria:

* SCID-confirmed (Structured Clinical Interview for DSM-IV Axis I Disorders) diagnosis of schizophrenia
* ages 18-55

Exclusion Criteria:

* history of substance abuse or dependence within 3 months; (ii) positive urine drug screen
* history or evidence of any disorder that might adversely influence cognitive measures (e.g. mental retardation)
* presence of serious neurological or general medical condition (e.g., Parkinson's disease, cardiac arrhythmia, epilepsy)
* clinical or laboratory evidence of uncompensated cardiovascular, endocrine, hematologic, hepatic, pulmonary (including bronchial asthma), or renal disease, narrow-angle glaucoma, malignant melanoma
* pregnancy/nursing or women of child-bearing age not on regular contraceptive therapy (effects of L-dopa unknown)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
SANS - Schedule for the Assessment of Negative Symptoms | 8 weeks

SECONDARY OUTCOMES:
MATRICS-Consensus Cognitive Battery | 8 weeks
BPRS - Brief Psychotic Rating Scale | 8 weeks
SAPS - Schedule for the Assessment of Positive Symptoms | 8 weeks
NIMH-MATRICS Brief Negative Symptoms Scale | 8 weeks
CGI-S - Clinical Global Impression - Severity Scale | 8 weeks
QLS - Quality of Life Scale | 8 weeks
CDS - Calgary Depression Scale | 8 weeks
SAS - Simpson Angus Scale for Extrapyramidal Symptoms | 8 weeks
BARS - Barnes Akathisia Rating Scales | 8 weeks
AIMS - Abnormal Involuntary Movement Scale | 8 weeks
UKU - Udvalg for Kliniske Undersogelses | 8 weeks
  Measures General Side Effects
LUNSERS - Liverpool University Neuroleptic Side-Effect Rating Scale | 8 weeks
BIS-11 - Barrett Impulsivity Scale | 8 weeks
Y-BOCS - Yale-Brown Obsessive Compulsive Scale | 8 weeks
DAI - Drug Attitude Inventory | 8 weeks
fMRI - Functional Magnetic Resonance Imaging | 8 weeks
  Changes in Regional Brain Activity
SWN - Subjective Well-Being on Neuroleptics Scale | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Remington, MD PhD FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre. — http://www.camh.net/research